CLINICAL TRIAL: NCT06153472
Title: Effectiveness of a Virtual Reality-Based Sensory Stimulation Intervention in Preventing Delirium in Intensive Care Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Liang Surui, Dr, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023K089
Record Dates: First submitted 2023-11-16; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Delirium; Intensive Care Unit; Randomised Controlled Trial
Keywords: delirium; intensive care unit; randomised controlled trial; sensory stimulation; virtual reality
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: 2
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-based sensory stimulation (Experimental): Participants in the experimental group will receive VR-based sensory stimulation.
  Interventions: Device: VR-based intervention
- Usual care (No Intervention): Participants in the control group will receive usual care.

INTERVENTIONS:
Device: VR-based intervention — The Virtual Reality-based sensory stimulation intervention will last for up to fourteen days, with all interventions administered by a research team. The primary outcomes will include delirium incidence, duration, and severity. The secondary outcomes will encompass patients' psychological well-being (post-traumatic stress disorder, sleep quality, and ICU memory), patients' clinical outcomes, and other outcomes (quality of life, independence, and cognitive function).
  Arms: VR-based sensory stimulation

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a VR-based sensory stimulation system in preventing ICU delirium in patients. The main questions it aims to answer are:

Is the VR-based sensory stimulation system more effective in preventing ICU delirium compared to usual care? Does VR sensory stimulation improve patient psychological well-being and clinical outcomes in the ICU?

Participants will:

Experimental Group:

Engage in VR-based sensory stimulation sessions involving visual or/and auditory stimulation.

Control Group:

Receive usual care without additional VR-based interventions.

Comparison:

Researchers will compare the outcomes between the experimental group (receiving VR-based sensory stimulation) and the control group (receiving usual care) to determine the effects of VR sensory stimulation on ICU delirium prevention, as well as its impact on patient psychological well-being and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients admitted to the study setting will be recruited if they are have: (1) ≥ 18 years, (2) the first time admitted to ICU and (3) a Richmond Agitation-Sedation Scale (RASS) score ≥-3

Exclusion Criteria:

* Patients will be excluded if they have: (1) been diagnosed with dementia, delirium or acute psychiatric illness at admission, (2) been diagnosed with end-stage cancer, (3) severe hearing impairment and cannot be corrected by hearing aids and (4) been admitted to ICU with radioactive material.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence, duration and severity | From the date of randomization and continues until either fourteen days have passed, the patient is discharged from the Intensive Care Unit (ICU), or the patient passes away from any cause, whichever comes first.
  Delirium incidence means the number of patients who are delirious and delirium duration means the number of days that a patient is delirious.

SECONDARY OUTCOMES:
Sleep quality | From the date of randomization and continues until either fourteen days have passed, the patient is discharged from the Intensive Care Unit (ICU), or the patient passes away from any cause, whichever comes first.
  The Richards-Campbell Sleep Questionnaire (RCSQ) is employed to assess the sleep quality of ICU patients.
Post Traumatic Stress Disorder | At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first.
  The 17-item PTSD Checklist (PCL) correspond to the DSM-III-R symptoms of PTSD and serves as a self-report scale for assessing PTSD
ICU memory | At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first.
  The ICU-Memory Tool (ICU-M) will be used to measure ICU patients' ICU experience
Patients' clinical outcomes | At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first.
  Medical outcomes will be extracted by the outcome assessor from the electronic health care system upon participants' discharge.
Participants' quality of life | Enrollement; At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first; through study completion, an average of 6 month
  The EuroQol- 5 Dimension (EQ-5D) will be used to assess the participants' quality of life.
Independence function | Enrollement; At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first; through study completion, an average of 6 month
  Motor-FIM (Functional Independence Measure) will be used to measure the independence function.
cognitive function | Enrollement; At either the end of the fourteen-day period or when the patient is discharged from the Intensive Care Unit (ICU), whichever comes first; through study completion, an average of 6 month
  Cognitive-FIM (Functional Independence Measure) will be used to measure the cognitive function.

REFERENCES:
- [Derived] Liang S, Liu Y, Wen T, Luo D, He M, Tian J. Effectiveness of a virtual reality-based sensory stimulation intervention in preventing delirium in intensive care units: a randomised-controlled trial protocol. BMJ Open. 2025 Jan 15;15(1):e083966. doi: 10.1136/bmjopen-2024-083966. PMID 39819916